CLINICAL TRIAL: NCT04105348
Title: The Association of Diabetes Mellitus and Inflammatory Bowel Disease
Brief Title: Diabetes Mellitus and Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MM Youssif, principal investigator, Assiut University
Other Study IDs: DM and IBD
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD with DM
  Interventions: Diagnostic Test: HbA1c
- IBD without DM
  Interventions: Diagnostic Test: HbA1c

INTERVENTIONS:
Diagnostic Test: HbA1c — patients with raised investigations will be included in group 1 patients with normal investigations will be included in group 2
  Other Names: fasting blood glucose; 2 hours postprandial blood glucose

SUMMARY:
Diabetes mellitus is a hyperglycemic metabolic disorder due to insulin deficiency or resistance at its receptors, leads to impaired glucose metabolism and multi-organ affection; (optic, peripheral neurological, cardiovascular and renal).

DETAILED DESCRIPTION:
Inflammatory bowel disease; (Crohn's disease and ulcerative colitis), is chronic relapsing inflammation in the gastrointestinal tract due to complex interactions among genetic, environmental, gut microbiome, and immunologic factors.

Inflammatory bowel disease treatment inhibits the abnormal inflammatory response to heal intestinal tissue, relieve the abdominal pain, the diarrhea and the fresh bleeding per rectum, also decreases the frequency of flare-ups and maintains remission.

Amino-salicylates and antibiotics are step I drugs act on the intestinal lining and on presented inflammatory masses.

Corticosteroids are step II drugs on failure of step I drugs for adequate control of the Inflammatory bowel disease and rapid relief of symptoms and inflammation.

The immune modifying agents as azathioprine and 6 mercaptopurine are step III drugs on failure of the steroids.

Biologic agents are anti Tumor necrotic factor agents (infliximab and adalimumab) and non anti Tumor necrotic factor agents (vedolizumab, ustekinumab and natalizumab).

Inflammatory bowel disease may have endocrinal and metabolic associations in the form of; lipid abnormalities and insulin resistance. Also, insulin resistance and hyperglycemia may be due to steroid use as steroid upgrades (hepatic gluconeogenesis, inhibition of glucose uptake in adipose tissue, and impairment of insulin action).

There is no epidemiological evidence that Inflammatory bowel disease is a definite risk factor for diabetes. In this study, the association of diabetes in patients with Inflammatory bowel disease will be determined.

ELIGIBILITY:
Inclusion Criteria:

- All patients with IBD admitted at EL-Raghy Assiut university hospital in the period of first of October 2019 to the end of September 2020 The diagnosis of DM is confirmed by high random blood glucose level more than 200mg/dl three times per day or high HbA1c more than 6.5%.

The diagnosis of IBD is confirmed by colonic biopsy results after colonoscopy.

Exclusion Criteria:

* Patients didn't do colonoscopy or didn't get biopsy or with normal colonoscopy and biopsy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: IBD clinic or Patients addmited at El raghy hospital in assiut university with IBD
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
effect of IBD on DM | on addmision
  patients with raised; HbA1c, fasting blood glucose, 2 hours postprandial blood glucose

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Background] Basso PJ, Fonseca MT, Bonfa G, Alves VB, Sales-Campos H, Nardini V, Cardoso CR. Association among genetic predisposition, gut microbiota, and host immune response in the etiopathogenesis of inflammatory bowel disease. Braz J Med Biol Res. 2014 Sep;47(9):727-37. doi: 10.1590/1414-431x20143932. Epub 2014 Jul 25. PMID 25075576
- [Background] Bernstein CN, Blanchard JF, Rawsthorne P, Yu N. The prevalence of extraintestinal diseases in inflammatory bowel disease: a population-based study. Am J Gastroenterol. 2001 Apr;96(4):1116-22. doi: 10.1111/j.1572-0241.2001.03756.x. PMID 11316157
- [Background] Tigas S, Tsatsoulis A. Endocrine and metabolic manifestations in inflammatory bowel disease. Ann Gastroenterol. 2012;25(1):37-44. PMID 24714153
- [Background] van Raalte DH, Ouwens DM, Diamant M. Novel insights into glucocorticoid-mediated diabetogenic effects: towards expansion of therapeutic options? Eur J Clin Invest. 2009 Feb;39(2):81-93. doi: 10.1111/j.1365-2362.2008.02067.x. PMID 19200161